CLINICAL TRIAL: NCT05765747
Title: A Randomized Controlled Clinical Trial of Effectiveness of Yunnan Baiyao in Improving Fracture Pain
Brief Title: Effectiveness of Yunnan Baiyao in Improving Fracture Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M2022860
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-02

CONDITIONS: Distal Radius Fracture
MeSH Terms: conditions — Wrist Fractures | interventions — yunnan baiyao; Celecoxib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yunnan Baiyao (Experimental): The Yunnan Baiyao group will be given 4 times a day, 2 capsules each time after morning, afternoon and evening meals and before going to bed. One capsule of Baoxianzi will be provided for the first time to be taken at the same time with Yunnan Baiyao Capsule, which will be given continuously for 2 weeks.
  Interventions: Drug: Yunnan Baiyao
- celecoxib (Active Comparator): The celecoxib group will be given 1 capsule twice a day after breakfast and dinner for 2 weeks.
  Interventions: Drug: Celecoxib 200mg

INTERVENTIONS:
Drug: Yunnan Baiyao — Yunnan Baiyao group will be given 4 times a day, 2 capsules each time after morning, afternoon and evening meals and before going to bed. One capsule of Baoxianzi will be provided for the first time to be taken at the same time with Yunnan Baiyao Capsule, which will be given continuously for 2 weeks.
  Arms: Yunnan Baiyao
Drug: Celecoxib 200mg — The celecoxib group will be given 1 capsule twice a day after breakfast and dinner for 2 weeks.
  Other Names: celecoxib
  Arms: celecoxib

SUMMARY:
This will be a randomized, controlled, non-inferiority designed clinical trial. 56 qualified subjects will be selected and allocated 1:1 to Yunnan Baiyao group and celecoxib group. Each subject will be treated for 2 weeks and observed for 12 weeks, which will be lasted for 14 weeks during the whole trial. Yunnan Baiyao group will be given 4 times a day, 2 capsules each time after morning, afternoon and evening meals and before going to bed. One capsule of Baoxianzi will be provided for the first time to be taken at the same time with Yunnan Baiyao Capsule, which will be given continuously for 2 weeks. The celecoxib group will be given 1 capsule twice a day after breakfast and dinner for 2 weeks.

DETAILED DESCRIPTION:
his will be a randomized, controlled, non-inferiority designed clinical trial. 56 qualified subjects will be selected and allocated 1:1 to Yunnan Baiyao group and celecoxib group. Each subject will be treated for 2 weeks and observed for 12 weeks, which will be lasted for 14 weeks during the whole trial. Yunnan Baiyao group will be given 4 times a day, 2 capsules each time after morning, afternoon and evening meals and before going to bed. One capsule of Baoxianzi will be provided for the first time to be taken at the same time with Yunnan Baiyao Capsule, which will be given continuously for 2 weeks. The celecoxib group will be given 1 capsule twice a day after breakfast and dinner for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. The age of the subject is 20-70 years old;
2. Patients with distal radius fractures (Colles fractures) ;
3. Conservative treatment (closed reduction and fixation) after fracture;
4. Willingness to participate in this study and sign the informed consent form (ICF).

Exclusion Criteria:

1. Pathological fractures such as multiple fractures and cancer;
2. Patients with a history of severe chronic disease, such as hypertension, coronary heart disease, diabetes, tuberculosis, etc.;
3. Patients with endocrine diseases unsuitable for inclusion or other related diseases affecting bone metabolism, such as thyroid diseases of clinical significance as hyperparathyroidism, parathyrometaplasia, Paget's disease, Cushing's syndrome, nephrotic rickets, osteomalacia, rheumatoid arthritis, gout, multiple myeloma, osteogenesis insufficiency, etc.;
4. Complicated with malignant tumor, mental illness and other diseases that doctors think may affect the test process;
5. Currently using bone metabolism regulation drugs, such as teripartide, bisphosphonate, etc.;
6. Had a history of chronic pain and used painkillers daily before enrollment; Nonsteroidal anti-inflammatory drugs, opioids, and physical therapy for pain relief within a week after fracture;
7. pregnant and lactating women;
8. Allergic to Yunnan Baiyao or any excipients and celecoxib, or suffering from contraindications or intolerance indicated by the test drug;
9. continuous use of antibiotics;
10. Patients with coagulation dysfunction, receiving anticoagulant therapy or taking antiplatelet aggregation drugs.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Change of VAS pain scores from baseline after administration | within 14 weeks
  Pain was measured using a VAS, where the amount of pain recorded ranged from 0 (no pain) to 100 (unbearable pain).

SECONDARY OUTCOMES:
The time for fracture healing | within 14 weeks
  The degree of fracture healing was evaluated by observing 4 layers of cortex (anteroposterior and lateral) on X-ray films and mRUST score
Changes from baseline in Procollagen I N-Terminal Propeptide (P1NP) | within 14 weeks
  Concentration determination of P1NP with unit of ng/mL
Changes from baseline in β-C-terminaltelopeptide of typeⅠcollagen (β-CTX) | within 14 weeks
  Concentration determination of β-CTX with unit of ng/mL
Changes from baseline in lumbar bone mineral density (BMD) | within 14 weeks
  Assessment of bone mineral density at the lumbar spine

CONTACTS AND LOCATIONS:
Overall Officials: Chunli Song, Pro., Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No